CLINICAL TRIAL: NCT04095910
Title: Evaluation of the Planet Nutrition Program on Obesity Parameters in Mexican Schoolchildren: Pilot Randomized ControlledTrial
Brief Title: Evaluation of the Planet Nutrition Program on Obesity Parameters in Mexican Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Full time professor, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPN01
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Childhood Obesity
Keywords: Prevention; Obesity; Childhood; School-based Program; Lifestyle; Nutrition Education
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planet Nutrition program (Experimental): multidisciplinary school- based program
  Interventions: Behavioral: Planet Nutrition program
- Control Group (No Intervention): Normal curricular classes

INTERVENTIONS:
Behavioral: Planet Nutrition program — 1. - Nutritional education sessions: The study team previously worked on the development of a handbook called "Planet Nutrition" which contains around 26 topics of nutrition and health. Interns from the Nutritional Sciences Degree of the University of Sonora implemented the sessions. 2 classes of 1 hour were given weekly, adding 18 sessions in total, during regular school hours. The program contemplates the establishment of different objectives.
  2. - Physical activity: The classes were designed and implemented by interns from the Bachelor of Physical Culture and Sport from the University of Sonora along with a teacher from the study team. 3 weekly sessions of 1 hour were provided. The activities were held on the schoolyard court during normal school hours, independent of the physical activity classes of the school.
  3. - Indirect family participation: Six information brochures with different nutrition and health topics were sent to parents.
  Arms: Planet Nutrition program

SUMMARY:
Obesity prevention programs in schools are essential to promoting healthy lifestyles. There are programs with positive effects on obesity parameters, but only a few of them have didactic material for its dissemination. In United States they have effective programs (with materials for their implementation) and some are already being implemented in different schools. In Mexico our study group has developed a program called "Planet Nutrition" that includes a manual.The main aim of this study is to evaluate the efficacy of the program "Planet Nutrition"-a nutrition education and behaviour change program- on BMI Z score in school children compared to a control group at 9 weeks. This pilot stud is a randomized controlled trial. The study will be conducted with 41 participants. The primary outcome was the change in the BMI Z score from baseline to 9 weeks. Secondary outcomes were the changes from baseline to 9 weeks in body fat percentage, waist circumference, systolic and diastolic blood pressure, consumption of healthy and unhealthy food, physical activity and sedentary lifestyle, cardiorespiratory capacity and nutrition knowledge. Additionally BMI Z score will be measured at 23 weeks, after the summer vacations. Considering evidence that this period could have a negative impact on children´s weight.

DETAILED DESCRIPTION:
Fifth grade students from a public elementary school in Hermosillo, Sonora, Mexico were invited to participate in the program. The nutritionist team of the study made the request face to face in the classrooms. A printed invitation was delivered to be given to schoolchildren parents, in addition to the informed consent and assent along with a data questionnaire. To be included children must be in fifth grade from the chosen school and be between 9 to 12 years old. The exclusion criteria were, having or develop a medical condition, taking medication or having an intervention that affects body weight, having a condition that prevents physical activity (cardiovascular, respiratory, muscular, osteoarticular, etc.) at baseline or during the study, and withdrawal of the consent informed

ELIGIBILITY:
Inclusion Criteria:

* Fifth grade students of the chosen school.
* Having 9 to 12 years old.

Exclusion Criteria:

* Having a condition, taking medication or carrying out an intervention that affects body weight.
* Condition that impede physical activity including cardiovascular, respiratory, muscular and bone condition.
* Withdrawal of informed consent and assent.
* Development of a health problem or taking medication with effect on body weight during the study.
* Participate in another intervention or treatment for obesity management during the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Change in BMI z score | Baseline to 9 weeks
  First, the weight and height of the children were measured with a SECA digital scale and a stadiometer (SECA 213). Then, the BMI z score was obtained using the WHO Anthro Plus software, where the values of weight, age, date of birth and sex were considered.

SECONDARY OUTCOMES:
Change in body fat | Baseline to 9 weeks
  A tetrapolar electrical bioimpedance method (BIE) was used to obtain the resistance and reactance values. The measurement was made with the BIE team, RJL Quantum II. To estimate the body fat percentage, a validated equation in Mexican children was used.
Change in waist circumference | Baseline to 9 weeks
  The measurement was taken at the umbilical scar level, with the participant standing and on the upper garment (due to the lack of privacy) using a non-stretch tape measure.
Change in the consumption of healthy and unhealthy food | Baseline to 9 weeks
  The questionnaire consists of 12 questions about the consumption of healthy foods (fruits, vegetables, cereals, legumes, animal source food, dairy, etc.) and unhealthy (sugary drinks, salty snacks, sweets, pastries, sausages, etc..). The frequency ranges from never to more than twice a day.
Change in auto-reported physical activity and sedentary activities | Baseline to 9 weeks
  It was measured by a validated questionnarie for schoolchildren which includes nine questions about the frequency and time spent in physical activity and sedentary activities during the week and weekend.
Change in nutrition knowledge | Baseline to 9 weeks
  To assess the learning in the nutritional education sessions, a questionnaire designed by the study team was used. It consisted of 32 questions about nutrition and health. The answers consisted by multiple choice with 4 subsections (A-D) and true or false choices.
Change in systolic and diastolic blood pressure | Baseline to 9 weeks
  A digital sphygmomanometer, model Omron HEM-907, was used. Two measurements were made to obtain an average value of systolic and diastolic blood pressure.
Change in cardiorespiratory capacity | Baseline to 9 weeks
  It was measured by the Course Navette test to estimate the maxium oxygen consumption (Vo2 Max).The participants traveled a distance of 20 meters round trips, at the rhythm of a recording sound. The test is in one minute stages and the speed increases (0.85 km / h to 0.5 km / h). The participants were stopping when they felt tired. The test was carried out by the physical activity team of the study.
Change in BMI Z score | 9 weeks to 21 weeks
  It will be measured returning from summer vacations, following the same method.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Gortmaker SL, Peterson K, Wiecha J, Sobol AM, Dixit S, Fox MK, Laird N. Reducing obesity via a school-based interdisciplinary intervention among youth: Planet Health. Arch Pediatr Adolesc Med. 1999 Apr;153(4):409-18. doi: 10.1001/archpedi.153.4.409. PMID 10201726
- [Background] Shamah Levy T, Morales Ruan C, Amaya Castellanos C, Salazar Coronel A, Jimenez Aguilar A, Mendez Gomez Humaran I. Effectiveness of a diet and physical activity promotion strategy on the prevention of obesity in Mexican school children. BMC Public Health. 2012 Mar 1;12:152. doi: 10.1186/1471-2458-12-152. PMID 22381137
- [Background] WHO. 2007. Growth Reference 5-19 years. BMI-for-age (5-19 years). https://www.who.int/growthref/en/
- [Background] Diaz-Zavala RG, Castro-Cantu MF, Valencia ME, Alvarez-Hernandez G, Haby MM, Esparza-Romero J. Effect of the Holiday Season on Weight Gain: A Narrative Review. J Obes. 2017;2017:2085136. doi: 10.1155/2017/2085136. Epub 2017 Jul 4. PMID 28744374
- [Background] Franckle R, Adler R, Davison K. Accelerated weight gain among children during summer versus school year and related racial/ethnic disparities: a systematic review. Prev Chronic Dis. 2014 Jun 12;11:E101. doi: 10.5888/pcd11.130355. PMID 24921899
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, et al; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017; 140(3):e20171904. Pediatrics. 2017 Dec;140(6):e20173035. doi: 10.1542/peds.2017-3035. No abstract available. PMID 29192011
- [Background] Brown T, Moore TH, Hooper L, Gao Y, Zayegh A, Ijaz S, Elwenspoek M, Foxen SC, Magee L, O'Malley C, Waters E, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2019 Jul 23;7(7):CD001871. doi: 10.1002/14651858.CD001871.pub4. PMID 31332776
- [Background] Leger LA, Mercier D, Gadoury C, Lambert J. The multistage 20 metre shuttle run test for aerobic fitness. J Sports Sci. 1988 Summer;6(2):93-101. doi: 10.1080/02640418808729800. PMID 3184250
- [Background] Ramirez E, Valencia ME, Bourges H, Espinosa T, Moya-Camarena SY, Salazar G, Aleman-Mateo H. Body composition prediction equations based on deuterium oxide dilution method in Mexican children: a national study. Eur J Clin Nutr. 2012 Oct;66(10):1099-103. doi: 10.1038/ejcn.2012.89. Epub 2012 Jul 18. PMID 22805494
- [Background] Currie C, Griebler R, Inchley J, Theunissen A, Molcho M, Samdal O, Dür W. 2010. Health Behaviour in School-aged Children (HBSC) Study Protocol: Background, Methodology and Mandatory items for the 2009/10 Survey. Edinburgh: CHRU & Vienna: LBIHPR.